CLINICAL TRIAL: NCT04532580
Title: Clinical Validation of Boneview for FDA Submission: Evaluation of the Ability of the Artificial Intelligence Software, Boneview, to Improve Physicians' and Radiologists' Performances in Detecting Fractures on Bone X-Rays Radiographs.
Brief Title: Clinical Validation of Boneview for FDA Submission
Status: Completed | Type: Observational
Sponsor: Gleamer (Industry)
Responsible Party: Sponsor
Other Study IDs: BCK-CEP
Record Dates: First submitted 2020-08-25; First posted 2020-08-31 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Fracture
Keywords: fracture; artificial intelligence; x-rays radiographs
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- AI- Aided performances
  Interventions: Device: Diagnosis of fracture on X-Ray Radiographs
- AI- Unaided performances
  Interventions: Device: Diagnosis of fracture on X-Ray Radiographs

INTERVENTIONS:
Device: Diagnosis of fracture on X-Ray Radiographs — Diagnosis of fracture on X-Ray Radiographs with and without the assistance of Boneview Software

SUMMARY:
The goal of this clinical validation is to assess comparative performances of physicians with and without the assistance of BoneView for the diagnosis of fractures on radiographs.

The performances are evaluated in terms of accuracy (primary endpoint with the pair specificity/sensitivity and the secondary endpoint PPV/NPV) and in terms of time needed for diagnosis (secondary endpoint with the measurement of time on each case).

ELIGIBILITY:
Inclusion Criteria:

* Anonymized standard X-ray exams of extremity/pelvis/rib cage/dorsolumbar spine not containing or containing fracture(s).
* Adult patient, with minimum age of 21 years old.

Exclusion Criteria:

* Exams with one or more images including a body part not concerned by the intended use of BoneView (skull and cervical spine)
* Cases with one or more images being used for model design and development.
* Exams with one or more images being of poor quality (lossy), which prevent a proper interpretation by the readers.
* Cases not containing a medically relevant number of views for correct diagnosis.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The cases are consecutively sampled considering (non-)inclusion criteria (see below), and following these constraints:
  * At least 60 exams for the foot/ankle region, 60 exams for the knee/leg region, 60 exams for the hip/pelvis region, 60 exams for the hand/wrist region, 60 exams for the elbow/arm region, 60 exams for the shoulder/clavicula region, 60 exams of the rib cage region, 60 exams of the dorsolumbar spine region
  * 50% of exams of each region being positive: namely presenting one or multiple fracture(s) and 50% of exams of each region being negative: namely presenting no fracture
  * 50% of positive exams of each anatomical region presenting at least a "non-obvious" fracture and 50% with only "obvious" fracture(s). The determination of the "obvious" and "non-obvious" nature of the fractures would be determined during the Ground Truth determination process. The two osteo-articular experts that are performing the Ground Truth have to state the nature of the fracture.
Sampling Method: Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
measurement of diagnosis performances via calculation of sensitivity, specificity, NPV, PPV | 1 month
  calculation of sensitivity, specificity, NPV, PPV and comparison between the two cohorts

SECONDARY OUTCOMES:
Time needed for diagnosis via measurement of the time before submission of the diagnosis | 1 month
  measurement of the time and comparison between the two cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Nor-Eddine Regnard, MD, Study Chair — Gleamer
Locations (1):
- Boston Imaging Core Lab, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
no sharing of our IPD